CLINICAL TRIAL: NCT05253963
Title: Acute Effect of Continuous Positive Airway Pressure (CPAP) on Weight in Patients With Previously Untreated Obstructive Sleep Apnea
Brief Title: Acute Effect of CPAP on Weight in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Rodrigues Genta, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: acuteweightgain
Record Dates: First submitted 2021-09-29; First posted 2022-02-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure; Weight Gain
MeSH Terms: conditions — Sleep Apnea, Obstructive; Weight Gain | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): During the first and second study nights, subjects will undergo baseline polysomnography.
- Continuous Positive Airway Pressure (Experimental): Baseline polysomnography will be perfomed during the first study night and CPAP titration polysomnography will be performed during the second study night.
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure will be used during the second night of polysomnography .
  Arms: Continuous Positive Airway Pressure

SUMMARY:
The effect of CPAP on weight and fluid homeostasis will be assessed. Obstructive sleep apnea treatment-naive subjects will randomized to CPAP and control groups. Weight change, and changes in overnight urinary volume, intra and extracelullar volume, plasmatic B-type natriuretic peptide (BNP) and antidiuretic hormone (ADH) and urinary osmolality will be compared between groups.

DETAILED DESCRIPTION:
There is a bidirectional relationship between Obstructive Sleep Apnea (OSA) and obesity. Although obesity can lead to OSA, patients with OSA are more likely to gain weight. The mechanisms that lead to weight gain during the treatment of OSA are not known. Some evidence supports the hypothesis that fluid accumulation could be a possible explanation for weight gain after treatment for OSA. The hypothesis is that one night of CPAP treatment promotes increased body weight and reduced diuresis in patients with OSA. Participants will be submitted to 2 consecutive nights of polysomnography (PSG). A baseline PSG will be performed during the first study visit. During the second study night, participants will be randomized into two groups, CPAP and control (repeat baseline PSG). Overnight urinary volume will be determined. Intra and extracellular water volume will be assessed using electrical bioimpedance before bedtime and just after the subject wakes up. Plasmatic BNP and ADH and urinary osmolality will also be determined during each morning following PSG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Obstructive Apnea Sleep
* Over 18 years of age
* No previous treatment with Continuous Positive Airway Pressure

Exclusion Criteria:

* Congestive heart failure
* Renal insufficiency
* Hepatic failure
* Urinary incontinency
* Diuretic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Weight change | After 6 hours of Continuous Positive Airway Pressure treatment
  Weight change with just one night of CPAP treatment.
Diuresis change | After 6 hours of Continuous Positive Airway Pressure treatment
  diuresis change with just one night of CPAP treatment.

SECONDARY OUTCOMES:
Urinary osmolarity | After 10 hours of the nocturnal polysomnography
  Urine will be collected
Atrial natriuretic peptide and antidiuretic hormone | After 10 hours of the nocturnal polysomnography
  Blood samples will be collected
Intra and extracellular fluid volume | Before the beginning and after 10 hours of the nocturnal polysomnography.
  Intra and extracellular fluid volume accumulation will be assessed by bioelectrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Pedro R Genta, MD.PhD, Principal Investigator — Sleep Laboratoy, Heart Institute
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lima GF, Herculano S, Fernandes MD, Lima-Junior JGA, Alves RSC, Drager LF, Lorenzi-Filho G, Genta PR. Acute Effect of Continuous Positive Airway Pressure (CPAP) on Weight in Patients with Obstructive Sleep Apnea: A Randomized Study. Ann Am Thorac Soc. 2025 Sep 30. doi: 10.1513/AnnalsATS.202505-491OC. Online ahead of print. PMID 41025888